CLINICAL TRIAL: NCT02988739
Title: Safety and Immunogenicity of Laser Assisted Epidermally Administered Seasonal Influenza Vaccine in Comparison to Intradermally Administered Seasonal Influenza Vaccine
Brief Title: Comparison of Laser Assisted Epidermal to Intradermal Administration of Seasonal Influenza Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pantec Biosolutions AG (Industry)
Collaborators: Medical University of Vienna (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PCT-007
Record Dates: First submitted 2016-12-06; First posted 2016-12-09 (Estimated); Last update posted 2018-03-06 (Actual); Status verified 2018-03

CONDITIONS: Influenza in Human
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser assisted epidermal application (Experimental): Laser pretreatment: 4 adjacent areas of 2 cm² each (14mm x 14 mm) will be pretreated with an Erbium Yttrium Aluminium Garnet laser (22,7 J/cm², 2 pulses, Density: 5%) generating micropores with a depth of approximately 91 µm.
  0,1 ml of Intanza (15 µg, seasonal trivalent influenza vaccine) will be topically administered on the laser-treated area.
  Interventions: Biological: seasonal influenza vaccine; Device: fractional Er:Yag laser
- Intradermal application (Active Comparator): 0,1 ml of Intanza (15 µg, seasonal trivalent influenza vaccine) will be intradermally injected in the deltoid area.
  Interventions: Biological: seasonal influenza vaccine

INTERVENTIONS:
Biological: seasonal influenza vaccine — influenza vaccine containing 15 µg haemagglutinin of three seasonal influenza virus strains recommended by WHO
  Other Names: INTANZA
Device: fractional Er:Yag laser — Fraction laser device to apply micorpores of defined depth and density into skin.
  Other Names: Pantec P.L.E.A.S.E.
  Arms: Laser assisted epidermal application

SUMMARY:
It is the aim of the present study to compare the immunogenicity induced by a laser-assisted epidermally administered seasonal influenza vaccine to an intradermally administered seasonal influenza vaccine.

DETAILED DESCRIPTION:
The skin is an attractive tissue for vaccination due to the impact of the cutaneous micro-environment on the adaptive and non-adaptive immune responses. Conventionally many vaccines are administered subcutaneously. Immune-competent cells however are not resident in the subcutaneous fat tissue, but instead are located in the epidermis and the dermis of the skin. Depending on the targeted skin layer and administration method, different immunological outcomes are thus anticipated following vaccination.

In the present study, the immunogenicity (in terms of activation of B-cell mediated and T-cell mediated immune responses) of laser-assisted epidermally administered seasonal influenza vaccine will be compared to needle-based intradermal administration of the same seasonal influenza vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* 18-30 years old (male or female),
* Photo type I to IV (according to Fitzpatrick scale),
* Subject must be willing and able to comply with study protocol for the duration of the study,
* Females of childbearing potential (FCB) must maintain reliable contraception throughout the study.

Exclusion Criteria:

* Known pregnancy or positive pregnancy test for women of child bearing potential,
* Positive screening assessment for human immunodeficiency virus or viral hepatitis (Hepatitis B or Hepatitis C)
* Known or suspected immune dysfunction that is caused by a medical condition, or any other cause and that would interfere with the conduct of the study,
* Use, within the past 3 months, of any topical or systemic treatment that would interfere with assessment and/or investigational treatment (anti-inflammatory drugs, immune suppressors or any immune modulator agent),
* Use of any topical treatment on the injection site within the last four weeks,
* Photo type V and VI (according to Fitzpatrick scale),
* Skin lesions or excessive hair growth at treatment site,
* Any history of seasonal influenza in the past 6 months,
* Any seasonal influenza vaccine in the past,
* Preexisting HAI antibody titers of >40 against more than one influenza strain included in the vaccine,
* Acute illness or febrile illness (over 37,5°C) within one week prior to enrollment,
* Hypersensitivity to elements of the influenza vaccine (e.g. egg),
* Administration of any live vaccine (< 28 days) or inactivated/toxoid vaccine (< 14 days) or planned vaccination within 3 months after inclusion,
* Medical history of skin cancer,
* History of Guillain Barre syndrome or brachial neuritis following previous vaccination,
* Any history of having blood transfusions or administration with gamma globulin in the past 3 months
* Women of childbearing potential not actively practicing birth control or using medically accepted device or therapy,
* Subject being judged as inadequate for following the procedures of the trial by investigator,
* Participation in another clinical trial (including follow up phase of a previous clinical trial)

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2017-02-22 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Haemagglutination inhibition (HAI) | day 1 and day 29
  HAI against each vaccine virus strain
Frequency of vaccine specific T-cell responders | day 1, day 15 and day 29
  Number of subjects achieving a T-cell stimulation index of >3

SECONDARY OUTCOMES:
Seroconversion rate | day 1 and day 29
  Proportion of subjects achieving at least a four fold HAI titer increase against each vaccine virus strain from day 1 to day 29
Seroprotection rate | day 1 and day 29
  Proportion of subjects achieving a HAI titer of > 1:40 against each vaccine virus strain at day 29
Geometric Mean fold rise (GMFR) of antibody titers | day 1 and day 29
  GMFR of antibody titers against each vaccine virus strain from day 1 to day 29.
Magnitude of T-cell response | day 1 , day 15 and day 29
  Magnitude of T-cell response (SI values) against influenza vaccine on day 1, day 15 and day 29.
Frequency and severity of local and systemic adverse events following vaccination | day 1 to day 29

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University Vienna, University Clinic for Clinical Pharmacology, Vienna, Austria